CLINICAL TRIAL: NCT01241877
Title: Astaxanthin Supplementation in Cyclists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Peter Res, MUMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 10-3-068
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Athletic Performance
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- astaxanthin (Experimental)
  Interventions: Dietary Supplement: astaxanthin
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: astaxanthin — astaxanthin
  Arms: astaxanthin
Dietary Supplement: placebo — placebo
  Arms: placebo

SUMMARY:
Background of the study:

Astaxanthin has been shown to be a powerfull anti-oxidant. Health benefits have been shown in animals and humans. Exercise enhancing effects have been shown in animals via enhancement of fat oxidation. We want to examine the effects of 4 weeks of astaxanthin supplementation on fat oxidation and cycling performance in trained cyclists

Objective of the study:

To test the hypothesis that 4 weeks supplementation with astaxanthin will improve fat oxidation and improve exercise performance in trained cyclists

Study design:

Double blind, placebo controlled study.

Study population:

Well trained cyclists between 18-30 years old

Intervention (if applicable):

astaxanthin (20 mg/day) or placebo for 4 weeks

Primary study parameters/outcome of the study:

performance on a time trial after 90 min steady state exercise.

Secundary study parameters/outcome of the study (if applicable):

substrate use plasma glucose plasma lactate plasma free fatty acid plasma astaxanthin

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

The risks involved in participating in this experiment are minimal. Astaxanthin has been shown to be safe. Insertion of the catheters in a vein is comparable to a normal blood draw and the only risk is of a small local haematoma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* Age between 18 and 30 years
* Endurance trained (≥3 sessions of endurance exercise per week)
* VO2 max ≥ 50 ml/kg/min
* Training history of more than one year of ≥3 sessions of endurance exercise per week
* BMI <25 kg/m2

Exclusion Criteria:

* Use of medication
* Smoking

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
time trial performance | 4 weeks
  time trial performance

SECONDARY OUTCOMES:
substrate use | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, LI, Netherlands

REFERENCES:
- [Derived] Klinkenberg LJ, Res PT, Haenen GR, Bast A, van Loon LJ, van Dieijen-Visser MP, Meex SJ. Effect of antioxidant supplementation on exercise-induced cardiac troponin release in cyclists: a randomized trial. PLoS One. 2013 Nov 19;8(11):e79280. doi: 10.1371/journal.pone.0079280. eCollection 2013. PMID 24260184